CLINICAL TRIAL: NCT02894216
Title: Clinical Value of Radionuclide Shuntography by Qualitative Methods in Hydrocephalic Adult Patients With Suspected Ventriculoperitoneal Shunt Malfunction
Brief Title: Qualitative Radionuclide Shuntography for Adult Patients With Suspected V-P Shunt Malfunction
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Szu-Ying Tsai, Resident doctor, Far Eastern Memorial Hospital
Other Study IDs: 105026-E
Record Dates: First submitted 2016-05-04; First posted 2016-09-09 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Ventriculoperitoneal Shunt Malfunction; Radionuclide Shuntography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: radionuclide shuntography — the investigators retrospectively enrolled patient who received radionuclide shuntography

SUMMARY:
The investigators retrospectively reviewed all radionuclide shuntographic tests using (99m)technetium-pertechnetate (DTPA) performed between August 2005 and December 2015 in nuclear medicine department of Far Eastern Memorial Hospital. The results of shuntography were evaluated visually and qualitatively, and correlated with clinical follow-up. The tests were interpreted as normal and abnormal, including complete distal obstruction, partial distal obstruction or miscellaneous. Clinical outcomes within 30 days were defined based on subsequent need for revision, re-implantation or adjustment of shunt pressure. Then the investigators calculated the sensitivity (Se), specificity (Sp), positive predictive value (PPV), negative predictive value (NPV) and overall accuracy.

DETAILED DESCRIPTION:
Introduction: Cerebrospinal fluid ventriculoperitoneal (V-P) shunts are often used in the treatment of hydrocephalus. Complications from shunts are not uncommon and can present with a variety of signs and symptoms, which could be evaluated by clinical examination and neuro-imaging. The radionuclide cerebrospinal fluid (CSF) shunt study provides a simple, effective, and low-radiation-dose method of assessing CSF shunt patency. When a discrepancy between neurological examination and imaging, additional radionuclide shuntography can be helpful. The purpose of the study was to analyze in the imaging findings and clinical interpretation of a variety of shuntography results and to determine the applicability of shuntography in patients with suspected shunt malfunction.

Materials and Methods: The investigators include all radionuclide shuntographic tests using (99m)technetium-pertechnetate (DTPA) performed between August 2005 and December 2015 in our department. No complications or discomfort were noted in the examinations. The results of shuntography were evaluated visually and qualitatively, and correlated with clinical follow-up. The tests were interpreted as normal and abnormal, including complete distal obstruction, partial distal obstruction or miscellaneous. Clinical outcomes within 30 days were defined based on subsequent need for revision, re-implantation or adjustment of shunt pressure. Then the investigators calculated the sensitivity (Se), specificity (Sp), positive predictive value (PPV), negative predictive value (NPV) and overall accuracy. The investigators would also determine the correlation with operative findings and assessment of radionuclide shuntography.

ELIGIBILITY:
Inclusion Criteria:

* all radionuclide shuntographic tests using (99m)technetium-pertechnetate (DTPA) performed between August 2005 and December 2015 in nuclear medicine department in Far Eastern Memorial Hospital

Exclusion Criteria:

* patients younger than 21 years old

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators include all radionuclide shuntographic tests using (99m)technetium-pertechnetate (DTPA) performed between August 2005 and December 2015 in our department. No complications or discomfort were noted in the examinations. The results of shuntography were evaluated visually and qualitatively, and correlated with clinical follow-up. The tests were interpreted as normal and abnormal, including complete distal obstruction, partial distal obstruction or miscellaneous. Clinical outcomes within 30 days were defined based on subsequent need for revision, re-implantation or adjustment of shunt pressure. Then the investigators calculated the sensitivity (Se), specificity (Sp), positive predictive value (PPV), negative predictive value (NPV) and overall accuracy. The investigators would also determine the correlation with operative findings and assessment of radionuclide shuntography.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
clinical outcome | 30 days post radionuclide shuntography
  subsequent need for revision, re-implantation or adjustment of shunt pressure.

SECONDARY OUTCOMES:
surgical findings | 30 days post radionuclide shuntography
  findings (obstruction or not) noted by surgery

OTHER OUTCOMES:
Safety and Tolerability - Number of participants with treatment-related adverse events | 30 days post radionuclide shuntography
  Number of participants with treatment-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Ying Tsai, MD, Principal Investigator — Far Eastern Memorial Hospital

IPD SHARING:
Plan to Share IPD: No